CLINICAL TRIAL: NCT03632876
Title: Vitamin A in Sickle Cell Disease: Improving Sub-optimal Status With Supplementation
Brief Title: Nutritional Outcomes After Vitamin A Supplementation in Subjects With SCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Penn State University (Other); Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-010081
Record Dates: First submitted 2018-08-01; First posted 2018-08-16 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Sickle Cell Anemia in Children; Vitamin A Deficiency in Children
Keywords: Retinol; Stable isotope dilution; DXA; retinyl palmitate
MeSH Terms: interventions — retinol palmitate

STUDY DESIGN:
Intervention Model Description: Subjects in parallel groups will be randomized to one of two doses of vitamin A supplementation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lower Dose Vitamin A (Active Comparator): Subjects with SCD-SS in the lower dose Vitamin A arm receive 3000IU of retinyl palmitate daily for 8 weeks.
  Interventions: Dietary Supplement: retinyl palmitate
- Higher Dose Vitamin A (Active Comparator): Subjects with SCD-SS in the higher dose Vitamin A arm receive 6000IU of retinyl palmitate daily for 8 weeks.
  Interventions: Dietary Supplement: retinyl palmitate
- Healthy Comparison Arm (No Intervention): Healthy subjects receive no intervention and undergo comparisons to the two vitamin A supplementation arms at baseline.

INTERVENTIONS:
Dietary Supplement: retinyl palmitate — The intervention is a daily vitamin A supplement.
  Arms: Higher Dose Vitamin A; Lower Dose Vitamin A

SUMMARY:
This study establishes the safety and efficacy of vit A supplementation doses (3000 and 6000 IU/d) over 8 weeks in children with SCD-SS, ages 9 and older and test the impact of vit A supplementation on key functional and clinical outcomes. Additionally, vitamin A status is assessed in healthy children ages 9 and older to compare to subjects with SCD-SS.

DETAILED DESCRIPTION:
Suboptimal vitamin A (vit A) status is prevalent in children with type SS sickle cell disease (SCD-SS) and associated with hospitalizations and poor growth and hematological status. Preliminary data in children with SCD-SS show that vit A supplementation at the dose recommended for healthy children failed to improve vit A status, resulting in no change in hospitalizations, growth or dark adaptation. This indicates an increased vit A requirement most likely due to chronic inflammation, low vit A intake and possible stool or urine loss. The dose of vit A needed to optimize vit A status in subjects with SCD-SS is unknown.

ELIGIBILITY:
Inclusion Criteria:

* Sickle cell disease, SS genotype (subjects with sickle cell disease only)
* Usual state of good health (no hospitalizations, emergency room visits, or unscheduled acute illness clinic visits for two weeks prior to screening)
* Commitment to a 119-day study (subjects with sickle cell disease only), or a 4-day study (healthy volunteers only)

Exclusion Criteria:

* Hydroxyurea initiated within the previous 6 weeks (subjects with sickle cell disease only)
* History of stroke (subjects with sickle cell disease only)
* Other chronic conditions that may affect growth, dietary intake or nutritional status
* Retinoic acid (topical or oral), weight loss medication and/or lipid lowering medications
* Subjects with a BMI greater than 98th percentile for age and sex
* Pregnant or lactating females (subjects who become pregnant during the course of the study will not continue participation)
* Liver function tests >4 x upper limit of reference range
* Participation in another study with impact on vitamin A status (subjects with sickle cell disease only)
* Use of multi-vitamin or commercial nutritional supplements containing vitamin A (those who are willing to discontinue these supplements, with the approval of the medical care team, will be eligible for the study after a 1 month washout period. Subjects taking nutritional products without vitamin A will be eligible)
* Inability to swallow pills (subjects with sickle cell disease only)

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-10-02 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Serum Vitamin A status | Change from baseline after supplementation for 8 weeks
  Serum vitamin A as measured by retinol

SECONDARY OUTCOMES:
Vitamin A toxicity | Change from baseline after supplementation for 8 weeks
  Retinyl palmitate
Height Z-score | Change from baseline after supplementation for 8 weeks
  Measured on a stadiometer, compared to Center for Disease Control (CDC) reference standard to create a z-score
Weight Z-score | Change from baseline after supplementation for 8 weeks
  Measured on a standing scale, compared to CDC reference standard to create a z-score
BMI Z-score | Change from baseline after supplementation for 8 weeks
  Calculated using kg/m^2 and compared to CDC reference standards
Fat-free Mass | Change from baseline after supplementation for 8 weeks
  Calculated from dual-energy x-ray absorptiometry (DEXA) scan
Fat-free Mass | Change from baseline after supplementation for 8 weeks
  Calculated from DEXA scan
Fat Mass | Change from baseline after supplementation for 8 weeks
  Calculated from DEXA scan
Upper arm muscle area | Change from baseline after supplementation for 8 weeks
  Calculated from mid-upper arm circumference
Upper arm fat area | Change from baseline after supplementation for 8 weeks
  Calculated from mid-upper arm circumference and triceps skinfold thickness
Muscle strength | Change from baseline after supplementation for 8 weeks
  Directly measured with Biodex Multi-Joint System 3 Pro
Jump strength | Change from baseline after supplementation for 8 weeks
  Directly measured with Force Plate
Upper limb strength | Change from baseline after supplementation for 8 weeks
  Directly measured with hand-grip strength dynamometer
Muscle function | Change from baseline after supplementation for 8 weeks
  Directly measured with Bruininks-Oseretsky Test of Motor Proficiency
Dietary Intake | Change from baseline after supplementation for 8 weeks
  Analysis of a three-day food record
Coefficient of fat absorption | Change from baseline after supplementation for 8 weeks
  Calculated from 72-hour stool collection and dietary fat intake
Hemoglobin | Change from baseline after supplementation for 8 weeks
  Direct measurement through spectral absorption
Hematocrit | Change from baseline after supplementation for 8 weeks
  Direct measurement through spectral absorption
Fetal hemoglobin | Change from baseline after supplementation for 8 weeks
  Direct measurement through quantitative flow cytometry
Mean corpuscular volume | Change from baseline after supplementation for 8 weeks
  Direct measurement through quantitative flow cytometry
Mean corpuscular hemoglobin | Change from baseline after supplementation for 8 weeks
  Calculated from hemoglobin mass and erythrocyte count
Mean corpuscular hemoglobin concentration | Change from baseline after supplementation for 8 weeks
  Calculated from hemoglobin divided by hematocrit
Reticulocyte count | Change from baseline after supplementation for 8 weeks
  Direct measurement through quantitative flow cytometry
Retinol binding protein, serum | Change from baseline after supplementation for 8 weeks
  Direct measurement through quantitative nephelometry
Retinol binding protein, urine | Change from baseline after supplementation for 8 weeks
  Direct measurement through quantitative nephelometry
Urine creatinine | Change from baseline after supplementation for 8 weeks
  Direct measurement through quantitative spectrophotometry
Serum creatinine | Change from baseline after supplementation for 8 weeks
  Direct measurement through quantitative spectrophotometry
Serum alanine aminotransferase | Change from baseline after supplementation for 8 weeks
  Direct measurement through quantitative enzymatic assay
Serum aspartate aminotransferase | Change from baseline after supplementation for 8 weeks
  Direct measurement through quantitative enzymatic assay
Serum gamma glutamyltransferase | Change from baseline after supplementation for 8 weeks
  Direct measurement through quantitative enzymatic assay
Serum alkaline phosphatase | Change from baseline after supplementation for 8 weeks
  Direct measurement through quantitative enzymatic assay
Serum bilirubin | Change from baseline after supplementation for 8 weeks
  Direct measurement through quantitative quantitative spectrophotometry
High-sensitivity c-reactive protein | Change from baseline after supplementation for 8 weeks
  Direct measurement through quantitative quantitative immunoturbidimetry
Tumor necrosis factor alpha | Change from baseline after supplementation for 8 weeks
  Direct measurement through quantitative quantitative multiplex bead assay
White blood cell count | Change from baseline after supplementation for 8 weeks
  Direct measurement through automated cell count
White blood cell differential | Change from baseline after supplementation for 8 weeks
  Direct measurement through automated cell count
Lymphocyte subtypes | Change from baseline after supplementation for 8 weeks
  Direct measurement through quantitative flow cytometry

OTHER OUTCOMES:
Total body vitamin A status via Stable Isotope Dilution | Change from baseline after supplementation for 8 weeks
  compartmental modeling of [13C10]-retinyl acetate, measured by high performance liquid chromatography/mass spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Stallings, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported will be shared upon request, after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be available immediately upon publication.
Access Criteria: Contact brownellj@email.chop.edu. Requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Ribaya-Mercado JD, Maramag CC, Tengco LW, Dolnikowski GG, Blumberg JB, Solon FS. Carotene-rich plant foods ingested with minimal dietary fat enhance the total-body vitamin A pool size in Filipino schoolchildren as assessed by stable-isotope-dilution methodology. Am J Clin Nutr. 2007 Apr;85(4):1041-9. doi: 10.1093/ajcn/85.4.1041. PMID 17413103
- [Background] Solomons NW. Vitamin A. In: B.Bowman, R.Russell, editors. Present Knowledge in Nutrition, Volume I. 9 ed. Washington DC: International Life Science Institute Press; 2006:157-183
- [Background] Ross CA. Vitamin A and carotenoids. In: M.E.Shils, M.Shike, C.A.Ross, B.Caballero, R.J.Cousins, editors. Modern Nutrition in Health and Disease. 10 ed. Philadelphia: Lippincott, Williams and Wilkins; 2006:351-375
- [Background] Schall JI, Zemel BS, Kawchak DA, Ohene-Frempong K, Stallings VA. Vitamin A status, hospitalizations, and other outcomes in young children with sickle cell disease. J Pediatr. 2004 Jul;145(1):99-106. doi: 10.1016/j.jpeds.2004.03.051. PMID 15238915
- [Background] Trumbo P, Yates AA, Schlicker S, Poos M. Dietary reference intakes: vitamin A, vitamin K, arsenic, boron, chromium, copper, iodine, iron, manganese, molybdenum, nickel, silicon, vanadium, and zinc. J Am Diet Assoc. 2001 Mar;101(3):294-301. doi: 10.1016/S0002-8223(01)00078-5. No abstract available. PMID 11269606
- [Background] Dougherty KA, Schall JI, Kawchak DA, Green MH, Ohene-Frempong K, Zemel BS, Stallings VA. No improvement in suboptimal vitamin A status with a randomized, double-blind, placebo-controlled trial of vitamin A supplementation in children with sickle cell disease. Am J Clin Nutr. 2012 Oct;96(4):932-40. doi: 10.3945/ajcn.112.035725. Epub 2012 Sep 5. PMID 22952182
- [Background] Haskell MJ, Handelman GJ, Peerson JM, Jones AD, Rabbi MA, Awal MA, Wahed MA, Mahalanabis D, Brown KH. Assessment of vitamin A status by the deuterated-retinol-dilution technique and comparison with hepatic vitamin A concentration in Bangladeshi surgical patients. Am J Clin Nutr. 1997 Jul;66(1):67-74. doi: 10.1093/ajcn/66.1.67. PMID 9209171
- [Background] Ribaya-Mercado JD, Solon FS, Solon MA, Cabal-Barza MA, Perfecto CS, Tang G, Solon JA, Fjeld CR, Russell RM. Bioconversion of plant carotenoids to vitamin A in Filipino school-aged children varies inversely with vitamin A status. Am J Clin Nutr. 2000 Aug;72(2):455-65. doi: 10.1093/ajcn/72.2.455. PMID 10919941
- [Background] Olson JA. Serum levels of vitamin A and carotenoids as reflectors of nutritional status. J Natl Cancer Inst. 1984 Dec;73(6):1439-44. PMID 6439934
- [Background] Kawchak DA, Schall JI, Zemel BS, Ohene-Frempong K, Stallings VA. Adequacy of dietary intake declines with age in children with sickle cell disease. J Am Diet Assoc. 2007 May;107(5):843-8. doi: 10.1016/j.jada.2007.02.015. PMID 17467383
- [Background] Garcia OP. Effect of vitamin A deficiency on the immune response in obesity. Proc Nutr Soc. 2012 May;71(2):290-7. doi: 10.1017/S0029665112000079. Epub 2012 Feb 28. PMID 22369848
- [Background] Cantorna MT, Nashold FE, Hayes CE. In vitamin A deficiency multiple mechanisms establish a regulatory T helper cell imbalance with excess Th1 and insufficient Th2 function. J Immunol. 1994 Feb 15;152(4):1515-22. PMID 8120366
- [Background] Esteban-Pretel G, Marin MP, Cabezuelo F, Moreno V, Renau-Piqueras J, Timoneda J, Barber T. Vitamin A deficiency increases protein catabolism and induces urea cycle enzymes in rats. J Nutr. 2010 Apr;140(4):792-8. doi: 10.3945/jn.109.119388. Epub 2010 Feb 24. PMID 20181784
- [Background] Kennedy KA, Porter T, Mehta V, Ryan SD, Price F, Peshdary V, Karamboulas C, Savage J, Drysdale TA, Li SC, Bennett SA, Skerjanc IS. Retinoic acid enhances skeletal muscle progenitor formation and bypasses inhibition by bone morphogenetic protein 4 but not dominant negative beta-catenin. BMC Biol. 2009 Oct 8;7:67. doi: 10.1186/1741-7007-7-67. PMID 19814781
- [Background] Dougherty KA, Schall JI, Rovner AJ, Stallings VA, Zemel BS. Attenuated maximal muscle strength and peak power in children with sickle cell disease. J Pediatr Hematol Oncol. 2011 Mar;33(2):93-7. doi: 10.1097/MPH.0b013e318200ef49. PMID 21228717
- [Background] Zemel BS, Kawchak DA, Ohene-Frempong K, Schall JI, Stallings VA. Effects of delayed pubertal development, nutritional status, and disease severity on longitudinal patterns of growth failure in children with sickle cell disease. Pediatr Res. 2007 May;61(5 Pt 1):607-13. doi: 10.1203/pdr.0b013e318045bdca. PMID 17413865
- [Background] Allen LH, Haskell M. Estimating the potential for vitamin A toxicity in women and young children. J Nutr. 2002 Sep;132(9 Suppl):2907S-2919S. doi: 10.1093/jn/132.9.2907S. PMID 12221269
- [Derived] Ford JL, Green MH, Brownell JN, Green JB, Oxley A, Lietz G, Schall JI, Stallings VA. Use of Compartmental Modeling and Retinol Isotope Dilution to Determine Vitamin A Stores in Young People with Sickle Cell Disease Before and After Vitamin A Supplementation. J Nutr. 2023 Sep;153(9):2762-2771. doi: 10.1016/j.tjnut.2023.07.004. Epub 2023 Jul 17. PMID 37468045